CLINICAL TRIAL: NCT02556970
Title: A Randomised Multi-centre Feasibility Study Investigating Post-operative Pain Following Single-port or Multi-port Video Assisted Thoracoscopic Surgical (VATS) Procedures
Brief Title: A Study Investigating Pain Following Single-port or Multi-port Video Assisted Thoracoscopic Surgery
Acronym: SiMuPort
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started and was abandoned.
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: David Telling Charitable Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU/2014/4744
Record Dates: First submitted 2015-09-04; First posted 2015-09-22 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Diclofenac; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-port surgery (Experimental): After induction of anaesthesia and lung isolation, a single intercostal incision will be placed laterally. This will usually be anterior to the border of the latissimus dorsi muscle, and in the 4th-7th space as appropriate to the planned surgery.
  A soft tissue wound protector can be used to protect the wound edges, but rigid intercostal retraction is not permitted. All instruments will be placed via this incision.
  Interventions: Procedure: Single port VATS; Drug: Paracetamol; Drug: Diclofenac; Device: Camera (5mm diameter 30 degree videothoracoscope); Device: Forceps grasper; Drug: 0.25% Levobupivicaine intercostal nerve block
- Multiple port surgery (Active Comparator): Patients in this arm will have 3 separate incisions placed to site the camera and other instruments. This will involve three separate incisions.
  Interventions: Drug: Paracetamol; Drug: Diclofenac; Device: Camera (5mm diameter 30 degree videothoracoscope); Device: Forceps grasper; Drug: 0.25% Levobupivicaine intercostal nerve block

INTERVENTIONS:
Procedure: Single port VATS — Performing video-assisted thorascopic surgery through a single port
  Arms: Single-port surgery
Drug: Paracetamol — 1g intraoperatively
  Other Names: Acetaminophen
Drug: Diclofenac — 75mg intraoperatively
  Other Names: Voltarol
Device: Camera (5mm diameter 30 degree videothoracoscope)
Device: Forceps grasper
Drug: 0.25% Levobupivicaine intercostal nerve block — Multi-level intercostal blocks will be placed subpleurally under thorascopic visualisation.
  Other Names: 0.25% Chirocaine

SUMMARY:
This study seeks to establish if thoracoscopic surgery performed through a single port or incision reduces early post-operative pain compared with conventional multiple port thoracoscopic surgery.

This initial pilot study is designed to establish whether a trial of the two techniques is acceptable to patients, clinically feasible and can be delivered in a reasonable timescale.

DETAILED DESCRIPTION:
This is a patient- and assessor-blinded, multi-centre randomised trial with two groups (n=20 in each arm). Patients referred to Universities Hospital Bristol NHS Foundation Trust (n=20) and Liverpool Heart and Chest Hospital NHS Foundation Trust (n=20) requiring elective VATS lung surgery.

Patients will be identified and recruited by the thoracic surgeons in their surgical outpatient clinic. Participants will receive verbal and written information about the two different surgical techniques.

Consent will be sought by one of the surgical research nurses in the surgical outpatient clinic after the thoracic surgeon has recruited them. On the rare occasion that this is not possible, consent will occur in the pre-operative assessment clinic (POAC) at a later date. All patients are seen in POAC at least 1 week prior to surgery except in extreme circumstances. In POAC consent will also be sought by one of the surgical research nurses.

Participants will be given contact details for the study team should they have any questions between consent and surgery. They will be able to withdraw consent at any time prior to surgery.

All data will be entered into a Trust-based computer that is password protected. Subject names will be kept on a database and will be linked only with a study identification number for this research. There will be no patient identifiers. Only the research team will have access to this computer. Data will be stored in a locked office and maintained for a minimum of five years after the completion of the study.

Participants will be block randomised 1:1 in blocks of 10 between single port surgery and multiple port surgery. Randomisation will occur by computer generation in theatre after induction of anaesthesia using the website www.sealedenvelope.com.

The treatment arm will involve performance of the planned surgical procedure through a single incision in the chest wall, without rib spreading. The camera and instruments will be placed through this single incision. Use of a soft tissue retractor is permitted.

The control arm will undergo the operation through a standard 3-incision approach, again without rib spreading.

All patients will receive skin dressings matching those for the multi-port technique, irrespective of randomised allocation. Patients will be informed not to remove these dressings for the first 24 hours. Surgical and anaesthetic staff members will be informed not to communicate information about the treatment allocation to the patient or nursing staff. The patient and the nursing staff undertaking pain assessments will not be aware of group allocation for the first 24 hours. The research nurses collecting the data will also be blinded.

The anaesthetic and surgical team involved cannot practically be blinded but will not be involved in outcome data collection.

All patients will receive simple intra-operative analgesia in the form of 1g intravenous paracetamol and 75mg intravenous diclofenac unless the patient is over 70 or has abnormal renal function. Extra opioid analgesia will be given as intravenous fentanyl or morphine and this will be titrated by the anaesthetist. The amount given will be documented as part of the trial data.

At the end of the procedure, multiple level (target at least 4) intercostal blocks will be placed subpleurally under thoracoscopic visualisation. 2ml of 2.5mg/ml Chirocaine (Levobupivicaine hydrochloride) will be injected into each space.

Post-operative analgesia will compromise of 1g paracetamol four times a day for the first 3 days after surgery. Patient will receive IV morphine titrated to pain in recovery and oramorph when they return to the ward. If patient is in significant pain a morphine patient controlled analgesia (PCA) will be set up in recovery and for the first night after surgery (1mg bolus, lockout 5mins). This will normally be discontinued on the first morning after surgery.

The following data will be recorded for all patients enrolled in the study:

Pre-operatively:

• At consent, a baseline quality of life score will be recorded.

Intra-operatively:

The following times will be recorded on a sticker attached to the patient's anaesthetic chart:

* Time of induction of anaesthesia
* Time of knife to skin
* Time of skin closure
* Time of extubation
* Time arrived in recovery These times will be recorded by the research nurses allowing the total surgical time (induction to skin closure) and total operative time (knife to skin to skin closure) to be calculated.

Post-operative period (expected to be 36-48 hours post-surgery):

* Visual Analogue Scale (VAS) pain scores are routinely recorded by the recovery nurses and ward nurses every hour for the first 24 hours post operatively and subsequently every 4 hours until discharge. So assuming the time into recovery is time zero the investigators will collect a pain score at time zero and then every hour for the first 24 hours. The investigators will then collect a pain score every 4 hours until discharge.
* Patient satisfaction survey will be conducted on day 1 and day 2 post-op.
* Total morphine consumption prior to discharge will be recorded.
* Time of discharge.
* Length of time chest drain remains in situ.
* Volume of blood loss in chest drain in first 24 hours.

At 30 days:

* All patients will complete a telephone quality of life score.
* Serious adverse events recorded in first 30 days:

  * Death
  * Readmission to hospital
  * Re-operation
  * Admission to ICU

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from patients requiring VATS for elective lung, lymph node or mediastinal biopsies or wedge resections of pulmonary nodules.
* Technically suitable for both single port or multiport approaches in the opinion of the recruiting surgeon.
* ASA 1,2 or 3.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Patient refusal.
* Emergency surgery.
* Patient unable to provide consent or complete the follow up.
* Patients who attend a chronic pain clinic on high doses of opiate drugs.
* History of Anaphylaxis/allergy to local anaesthetic.
* Lobectomy patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Ability to randomise 40 patients into trial | 3 months

SECONDARY OUTCOMES:
Median postoperative Visual Analogue Scale (VAS) pain score | Before discharge (24-48 hours)
  VAS pain score; 0 = no pain, 10 = worst pain participant could imagine
Maximum post operative Visual Analogue Scale (VAS) pain score | Before discharge (24-48 hours)
  VAS pain score; 0 = no pain, 10 = worst pain participant could imagine
Mean Visual Analogue Scale (VAS) pain score at 1 hour | 1 hour after surgery
  VAS pain score; 0 = no pain, 10 = worst pain participant could imagine
Mean Visual Analogue Scale (VAS) pain score at 24 hours | At 24 hours after surgery
  VAS pain score; 0 = no pain, 10 = worst pain participant could imagine
Crossover after randomisation | During surgery (normal surgical time is approximately 1 hour)
  Proportion of the trial (single port) arm converted to multiple port thoracoscopic or open approaches after randomisation
Total post-operative morphine consumption (mg) | In the first 24 hours post-surgery
  Total morphine dose in milligrams
Mortality | 30 days post-surgery
Unexpected ICU admission | After surgery and before discharge (expected to be with in 48 hours)
Hospital readmission rate | Within 30 days of surgery
  Readmission for any complication of the thoracic surgery.
Surgical site infection | Within 30 days of surgery
  Diagnosed infection in or around the surgical incisions.
Change in Quality of Life score | Performed pre-operatively and at 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Leslie, BM BS, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust